CLINICAL TRIAL: NCT03727594
Title: Radioguided Selective Neck Dissection for Staging and Treatment of Oral Cavity and Oropharyngeal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Nicola Malagutti, Principal Investigator, University Hospital of Ferrara
Other Study IDs: 151099
Record Dates: First submitted 2018-07-08; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to assess the role of lymphoscintigraphy as a simple and widely accessible method with a favorable cost/benefit ratio in improving oral cavity and oropharyngeal squamous cell carcinoma staging and surgical appropriateness and implementing a tailored surgical approach to cervical lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* accepted informed consent
* preoperative histological diagnosis of oral cavity or oropharyngeal squamous cell carcinoma
* patients fit to surgery of the primitive tumor and neck dissection (according to the general health condition and the clinical tumor stage)

Exclusion Criteria:

* rejected informed consent
* patients not fit to surgery (according to the general health condition and the clinical tumor stage)
* pregnant women

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by oral cavity or oropharyngeal squamous cell carcinoma admitted to our clinic.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with atypical lymphatic drainage of oral cavity and oropharyngeal squamous cell carcinoma identified through lymphoscintigraphy | 5 years
Number of metastasis or micrometastasis in the "sentinel" lymphnodes identified through immunofluorescence analysis of pancytokeratins | 5 years
Overall survival | 5 years
  Prognosis of radioguided neck dissection surgery compared to the standardized neck dissection traditionally performed in consideration of the site and the characteristics of the tumor and the clinical status of lymphnodes.
Disease-free survival | 5 years
  Prognosis of radioguided neck dissection surgery compared to the standardized neck dissection traditionally performed in consideration of the site and the characteristics of the tumor and the clinical status of lymphnodes.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy